CLINICAL TRIAL: NCT00249366
Title: Acute Drug Withdrawal in a General Medical Setting
Brief Title: Treatment of Alcohol Withdrawal in Hospital Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIAAAWEA-K2300222-A; K23AA000222 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Alcohol Withdrawal Syndrome
Keywords: Alcohol withdrawal; Symptom-triggered therapy; Fixed-schedule therapy; CIWA-Ar; Lorazepam (drug)
MeSH Terms: interventions — Lorazepam; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed-schedule treatment (Active Comparator): Fixed-schedule administration of lorazepam for alcohol withdrawal
  Interventions: Drug: Lorazepam (drug); Drug: Lorazepam
- Symptom-triggered treatment (Active Comparator): Symptom-triggered administration of lorazepam per protocol using the Clinical Institute Withdrawal Assessment for Alcohol, revised version (CIWA-Ar)
  Interventions: Drug: Lorazepam (drug); Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam (drug) — Lorazepam administered orally or IV for treatment of alcohol withdrawal in hospitalized patients
  Other Names: Ativan
Drug: Lorazepam — Lorazepam administered orally or IV for treatment of alcohol withdrawal in hospitalized patients
  Other Names: Ativan

SUMMARY:
The purpose of this study is to test how tolerable and effective lorazepam is when used to treat alcohol withdrawal in hospital patients at risk for alcohol withdrawal.

DETAILED DESCRIPTION:
Studies show that symptom-triggered dosing is best for treatment of alcohol withdrawal in patients on chemical dependence units without other illness. On general medical hospital wards, withdrawal may be affected by comorbid medical illness. A clinical trial was undertaken to determine whether there is a difference between symptom-triggered (ST) and fixed-schedule (FS) dosing of lorazepam in patients hospitalized on general medical wards at a University medical center. Subjects were assessed by their nurses with the Revised Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scale. Subjects in the ST arm received lorazepam doses based on CIWA-Ar score. Subjects in the FS arm received scheduled lorazepam with tapering over 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependence (based on criteria from the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition)
* Daily alcohol use for at least seven consecutive days with the last use no more than 72 hours prior to enrollment
* Patients on the General Internal Medicine service

Exclusion Criteria:

* Unable to give informed consent
* Chronically maintained on prescription sedative-hypnotics

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2001-04; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Withdrawal Assessment Scores | participants were followed for the duration of hospital stay, the median length of stay was 3 days
  Difference in Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scores between study arms
Total Dose of Lorazepam | participants were followed for the duration of hospital stay, the median length of stay was 3 days
  Differences in total amount of lorazepam administered between protocol groups
Protocol Errors | participants were followed for the duration of hospital stay, the median length of stay was 3 days
  Percentage of protocol errors between study arms, such as administration of an inappropriate lorazepam dose (inconsistent with CIWA-Ar score); excluded complications due to comorbid medical conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Weaver, MD, Principal Investigator — Virginia Commonwealth University Medical Center
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Result] Weaver MF, Hoffman HJ, Johnson RE, Mauck K. Alcohol withdrawal pharmacotherapy for inpatients with medical comorbidity. J Addict Dis. 2006;25(2):17-24. doi: 10.1300/j069v25n02_03. PMID 16785215